CLINICAL TRIAL: NCT06754462
Title: A Phase 2b, Multicenter, Double-blind, Placebo-controlled Randomized Withdrawal Study to Assess the Efficacy, Safety, and Tolerability of IMVT-1402 in Adult Participants With Active, Difficult to Treat, ACPA-Positive Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of IMVT-1402 in Adult Participants With Active, Difficult to Treat Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMVT-1402-2601; 2024-515973-82-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-24; First posted 2024-12-31 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anticitrullinated protein autoantibodies; Difficult-to-treat; Anti-FcRn; IMVT-1402; Autoimmune Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IMVT-1402 Dose 1 (Experimental)
  Interventions: Drug: IMVT-1402
- IMVT-1402 Dose 2 (Experimental)
  Interventions: Drug: IMVT-1402
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMVT-1402 — Administered once weekly by subcutaneous injection.
  Arms: IMVT-1402 Dose 1; IMVT-1402 Dose 2
Drug: Placebo — Administered once weekly by subcutaneous injection.
  Arms: Placebo

SUMMARY:
This Phase 2b, multicenter, double-blind, placebo-controlled, randomized withdrawal study is designed to assess the efficacy and safety of IMVT-1402 in adult participants with active, difficult-to-treat, anti-citrullinated protein autoantibody (ACPA) positive rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The primary objective is to evaluate the effects of IMVT-1402 compared to placebo, as measured by the American College of Rheumatology 20% (ACR20) response at Week 28.

The total duration of study participation is expected to be up to 86 weeks for an individual participant with 16 weeks of open-label treatment, 12 weeks of blinded randomized treatment, and 48 weeks of optional long-term extension treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants of age >18 years will be enrolled.
* Diagnosis of 'definite RA' according to the 2010 ACR/ European Alliance of Associations for Rheumatology (EULAR) Rheumatoid Arthritis Classification Criteria.
* Greater than or equal to 6/68 in tender joint count (TJC) and ≥ 6/66 swollen joint count (SJC) at both Screening and Baseline visits.
* C-reactive protein ≥ upper limit of normal (ULN) at Screening Visit.
* Elevated immunoglobulin G (IgG) + ACPA at the Screening Visit.
* Inadequate response to at least 2 classes of biologic/targeted synthetic disease-modifying antirheumatic drugs (DMARDs).

Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have received rituximab and experienced insufficient efficacy or loss of efficacy
* History of any chronic inflammatory arthritis with onset prior to age 18 or history of acute inflammatory joint disease of different origin from RA.
* Active malignancy or history of malignancy within 5 years prior to Screening Visit.
* Medical history of primary immunodeficiency, T cell or humoral, including common variable immunodeficiency.
* Used any nonimmunosuppressive fragment crystallizable (Fc)-based therapeutic protein (e.g., monoclonal antibody [mAb] or Fc-fusion protein) within 4 weeks prior to or at Screening Visit.
* Used any anti-FcRn treatment within 2 months prior to or at Screening Visit or have a documented history of non-response to prior anti-FcRn treatment.

Other, more specific exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who maintain ACR20 response at Week 28 | Week 28

SECONDARY OUTCOMES:
Change in Clinical Disease Activity Index (CDAI) score from Week 16 to Week 28 | Week 16 to Week 28
Change in Simplified Disease Activity Index (SDAI) score from Week 16 to Week 28 | Week 16 to Week 28

CONTACTS AND LOCATIONS:
Locations (83):
- United States (34):
  - Site Number - 1018, Mesa, Arizona
  - Site Number - 1019, Sun City, Arizona
  - Site Number - 1022, Covina, California
  - Site Number - 1028, San Leandro, California
  - Site Number - 1024, Temecula, California
  - Site Number - 1033, Tujunga, California
  - Site Number - 1023, Whittier, California
  - Site Number - 1020, Denver, Colorado
  - Site Number - 1015, Jupiter, Florida
  - Site Number - 1002, Miami, Florida
  - Site Number - 1027, Plantation, Florida
  - Site Number - 1005, Winter Park, Florida
  - Site Number - 1012, Zephyrhills, Florida
  - Site Number - 1001, Gainesville, Georgia
  - Site Number - 1034, Chicago, Illinois
  - Site Number - 1006, Cumberland, Maryland
  - Site Number - 1007, Hagerstown, Maryland
  - Site Number - 1031, Rockville, Maryland
  - Site Number - 1008, Worcester, Massachusetts
  - Site Number - 1021, Saint Clair Shores, Michigan
  - Site Number - 1030, Kansas City, Missouri
  - Site Number - 1010, Summit, New Jersey
  - Site Number - 1004, Charlotte, North Carolina
  - Site Number - 1035, Statesville, North Carolina
  - Site Number - 1000, Duncansville, Pennsylvania
  - Site Number - 1016, Jackson, Tennessee
  - Site Number - 1026, Memphis, Tennessee
  - Site Number - 1029, Murfreesboro, Tennessee
  - Site Number - 1037, Allen, Texas
  - Site Number - 1017, Colleyville, Texas
  - Site Number - 1036, Katy, Texas
  - Site Number - 1014, Mesquite, Texas
  - Site Number - 1013, Tomball, Texas
  - Site Number - 1025, Tomball, Texas
- Argentina (6):
  - Site Number - 5003, Buenos Aires
  - Site Number - 5001, Buenos Aires
  - Site Number -5004, Buenos Aires
  - Site Number - 5002, Buenos Aires
  - Site Number - 5005, Buenos Aires
  - Site Number - 5000, San Miguel de Tucumán
- Bulgaria (7):
  - Site Number - 5603, Plovdiv
  - Site Number - 5605, Plovdiv
  - Site Number - 5602, Plovdiv
  - Site Number - 5604, Rousse
  - Site Number - 5606, Sevlievo
  - Site Number - 5600, Sofia
  - Site Number - 5601, Sofia
- Czechia (5):
  - Site Number - 3204, Brno
  - Site Number - 3202, Ostrava
  - Site Number - 3203, Praha 2 Nove Mesto
  - Site Number - 3201, Uherské Hradiště
  - Site Number - 3200, Zlín
- Georgia (3):
  - Site Number - 8000, Tbilisi
  - Site Number - 8001, Tbilisi
  - Site Number - 8003, Tbilisi
- Germany (2):
  - Site Number - 6500, Hamburg
  - Site Number - 6501, Ratingen
- Hungary (6):
  - Site Number - 7554, Budapest
  - Site Number - 7555, Budapest
  - Site Number - 7550, Hódmezővásárhely
  - Site Number - 7553, Kecskemét
  - Site Number - 7551, Székesfehérvár
  - Site Number - 7552, Veszprém
- Poland (9):
  - Site Number - 3005, Bialystok
  - Site Number - 3007, Elblag
  - Site Number - 3009, Lublin
  - Site Number - 3006, Nadarzyn
  - Site Number - 3008, Poznan
  - Site Number - 3000, Poznan
  - Site Number - 3003, Sochaczew
  - Site Number - 3004, Warsaw
  - Site Number - 3002, Wroclaw
- Romania (3):
  - Site Number - 7500, Brasov
  - Site Number - 7502, Bucharest
  - Site Number - 7501, Râmnicu Vâlcea
- Spain (4):
  - Site Number - 7104, Barcelona
  - Site Number - 7101, Bilbao
  - Site Number - 7102, Málaga
  - Site Number - 7100, Seville
- United Kingdom (4):
  - Site Number - 7000, Edinburgh
  - Site Number - 7001, London
  - Site Number -7002, North Shields
  - Site Number - 7003, Wolverhampton

IPD SHARING:
Plan to Share IPD: No